CLINICAL TRIAL: NCT05444790
Title: Clinical Performance of NxTekTM Malaria P.f Plus Rapid Diagnostic Test Device and NxTekTM Malaria P.f/P.v Plus Rapid Diagnostic Test Device for the Detection of Plasmodium Infections in Patients With Symptoms Suggestive of Malaria for WHO Prequalification
Brief Title: Abbott NxTekTM Malaria RDT WHO Prequalification Study
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: University of Khartoum (Other); Eijkman Institute for Molecular Biology (Other); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Other Study IDs: MA016 Abbott
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Malaria; RDT; Diagnoses Disease
Keywords: Malaria, Diagnostics, RDT
MeSH Terms: conditions — Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid Diagnostic Test — The performance of two index tests and two comparator tests will be compared to reference tests and gold standard microscopy.
  Other Names: NxTekTM

SUMMARY:
Since their introduction in the late 90's, rapid diagnostic tests (RDTs) have dramatically improved our ability to control malaria but proved insufficient to support elimination efforts because of their limited sensitivity, especially for P. vivax. In addition, the spread of P. falciparum parasites lacking hrp2 gene jeopardizes the long-term use of P. falciparum-specific HRP2-based RDTs. A partnership between Abbott, FIND, PATH, and the Bill and Melinda Gates Foundation (BMGF) is addressing these limitations by developing two novel malaria RDTs with improved pLDH detection: a P. falciparum-specific test targeting both the HRP2 and PfLDH antigens on a single test line (NxTekTM Malaria P.f plus Rapid Diagnostic Test Device), and a P. falciparum/P. vivax combo test additionally targeting the PvLDH antigen on a second test line (NxTekTM Malaria P.f/P.v. plus Rapid Diagnostic Test Device).

These new combo tests with improved pLDH detection may provide added value compared to currently available malaria RDTs, especially in settings where current tests prove to be insufficient due to hrp2 deletion or high burden of P. vivax malaria.

Abbott, PATH, and FIND will conduct a prospective evaluation of NxTekTM Malaria P.f plus and NxTekTM Malaria P.f/P.v plus RDTs in malaria-endemic countries to assess their clinical performance for detection of malaria and usability in their intended-use settings. This is in support of a submission for WHO Prequalification.The purpose of this synopsis is to describe key points of alignment in study design and conduct across the portfolio of studies.

DETAILED DESCRIPTION:
Malaria continues to create a major health burden in the tropics especially in Africa. Introduction of Artemisinin-based combination therapy (ACT) has dramatically improved the outcomes of morbidity and mortality of malaria cases. Introduction of RDTs as well dramatically influenced cases detection hence treatment. The situation in Sudan is not different from the general picture in all Africa and witness great reduction of deaths from malaria since the introduction of ACT in 2005. The national protocol depends now on Giemsa stained slides microcopy or certified RDTs for diagnosis and ACT as first and second line of treatment.

Recommendation by World Health Organization (WHO) on parasitological confirmation of malaria cases by microscopy or rapid diagnostic tests (RDTs) before treatment increased the use and availability of RDTs worldwide.

Rapid diagnostic tests, since their introduction in the late 90's, have dramatically improved our ability to control malaria. Most RDTs are based on histidine-rich protein 2 (PfHRP2) or lactate dehydrogenase (pLDH), which are present in Plasmodium falciparum only and all human-infecting Plasmodium species respectively. However, the gradual spread of hrp2/hrp3-deleted mutants in several endemic countries in South America, Asia and Africa exerts a substantial potential impact on the utility of HRP2-based RDTs for case management in these settings.

Plasmodium lactate dehydrogenase (pLDH), on the other hand, appears as a good alternative to HRP2 as it is an essential protein expressed by all human-infecting Plasmodium species; however, pLDH-based RDTs were shown to perform poorly at low parasitaemia, which is common among patients infected with P. vivax, P. malariae and P. ovale species as well as in asymptomatic infections. Therefore, it is less preferred in endemic-countries. In these settings, malaria microscopy holds its reign as the standard of reference thanks to its low direct cost and ability to detect, quantify, and differentiate malaria parasites. However, it is also labour-intensive, time-consuming and expertise-demanding.

With the aim of addressing these limitations, Abbott has developed novel malaria RDTs, namely; NxTekTM Malaria Pf/Pv Plus and NxTekTM Malaria Pf Plus. These may provide added value compared to currently available malaria RDTs, especially in settings where current tests prove to be insufficient due to hrp2 deletion or high burden of P. vivax malaria.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years old or older
* Presenting at the study site with fever or a history of fever during the preceding 48 hours
* Freely agreeing to participate by providing informed consent (and assent, if applicable)

Exclusion Criteria:

* Presence of symptoms and signs of severe illness and/or central nervous system infections as defined by WHO guidelines

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms suggestive of malaria seeking clinical care in health facilities. By default, all such patients will be assessed for eligibility and, if appropriate, recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4563 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Point estimates of NxTekTM Malaria Pf Plus | 8 Months
  Point estimates of diagnostic accuracy characteristics (sensitivity, specificity, NPV, PPV) with 95% confidence intervals for NxTekTM Malaria Pf Plus using the reference test (nPCR) as standard of truth for the detection of P. falciparum infections in patients with symptoms suggestive of malaria.
Point estimates of NxTekTM Malaria Pf/Pv Plus | 8 Months
  Point estimates of diagnostic accuracy characteristics (sensitivity, specificity, NPV, PPV) with 95% confidence intervals for NxTekTM Malaria Pf/Pv Plus using the reference test as standard of truth for the detection of P. falciparum and P.vivax infections in patients with symptoms suggestive of malaria.

SECONDARY OUTCOMES:
Point estimates of comparator tests | 8 months
  Point estimates of diagnostic accuracy characteristics (sensitivity, specificity, NPV, PPV) with 95% confidence intervals of comparator tests using the reference test as standard of truth for the detection of P. falciparum and, P.vivax infections in patients with symptoms suggestive of malaria
Point estimates of index tests | 8 months
  Point estimates of diagnostic accuracy characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV) of the index tests for the detection of P. falciparum infections with hrp2 and/or hrp3 deletions in patients with symptoms suggestive of malaria.
User ability to read and interpret test | 8 months
  2.4 Percent of end users who can accurately interpret the investigational device result output.

CONTACTS AND LOCATIONS:
Locations (3):
- Exeins Health Institute, Jakarta, Indonesia
- Universidad Peruana Cayetano Heredia, Lima, Peru
- Institute of Endemic Diseases, Medical Campus, Khartoum, Sudan